CLINICAL TRIAL: NCT02172144
Title: A Double-blind, Randomised, Placebo Controlled, Six-way Crossover Study Including an Open-label Positive Control (Moxifloxacin) to Assess the Influence of Via Respimat® Inhaled BI 1744 CL (Single Doses of 10 μg, 20 μg, 30 μg and 50 μg) on the QT/QTc Interval of the ECG in Healthy Male and Female Volunteers
Brief Title: Via Respimat® Inhaled BI 1744 CL Compared to Moxifloxacin and Placebo in Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1222.8
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — Solutions; Inhalation; Moxifloxacin

ARMS (3):
- BI 1744 CL (Experimental)
  Interventions: Drug: BI 1744 CL solution for inhalation
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo matching BI 1744 CL
- Moxifloxacin (Avalox®) (Active Comparator)
  Interventions: Drug: Moxifloxacin (Avalox®)

INTERVENTIONS:
Drug: BI 1744 CL solution for inhalation
  Arms: BI 1744 CL
Drug: Placebo matching BI 1744 CL
  Arms: Placebo
Drug: Moxifloxacin (Avalox®)
  Arms: Moxifloxacin (Avalox®)

SUMMARY:
Study to investigate the effect of BI 1744 CL on the QT/QTc interval of the ECG (electrocardiogram) in comparison to placebo

ELIGIBILITY:
Inclusion Criteria:

All participants in the study will be healthy males or females, ranging from 21 to 50 years of age, with a body mass index (BMI) be within 18.5 to 29.9 kg/m2 (BMI calculation: weight in kilograms divided by the square of height in meters). In accordance with Good Clinical Practice and the local legislation all volunteers will have given their written informed consent prior to admission to the study

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders, clinically relevant electrolyte disturbances
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or clinically relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24:00 hours) within at least one month or less than ten half-lives of the respective drug before enrolment in the study or during the study
* Use of any drugs which might influence the results of the trial up to 7 days prior to enrolment in the study or during the study
* Participation in another trial with an investigational drug (within two months prior to administration or during the trial)
* Smoker (> 10 cigarettes or > 3 cigars of > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (> 60 g/day for males and > 20 g/day for females)
* Drug abuse
* Blood donation (> 100 mL within four weeks prior to administration or during the trial)
* Any laboratory value outside the reference range if indicative of underlying disease or poor health
* Excessive physical activities within the last week before the trial or during the trial
* Hypersensitivity to treatment medication, moxifloxacin and/or related drugs of these classes
* Previous tendon disease related to quinolone treatment
* Congenital or documented acquired QT- prolongation, previous history of symptomatic arrhythmias
* Pulse rate at screening of > 80 bpm or < 45 bpm
* Any screening ECG value outside of the reference range of clinical relevance including, but not limited to PR (Pulse rate) interval > 220 ms, QRS interval > 115 ms, QTcB > 450 ms, or QT (uncorrected) > 470 ms

For Female Subjects:

* Pregnancy
* Positive pregnancy test
* No adequate contraception (adequate contraception e.g. sterilisation, intrauterine-pressure, oral contraceptives)
* Inability to maintain this adequate contraception during the whole study period
* Lactation period

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2007-06; Primary Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the mean time-matched QTcI (QT interval, individually corrected according to the factor estimated from each subject) | Baseline (day -1) and 20 to 120 min. after drug administration

SECONDARY OUTCOMES:
Change of the QTcI at different point | Baseline (day -1) and 10 min. to 8 hours after drug administration
The mean of the QTcI values of all ECGs for Moxifloxacin and Placebo | 1 to 4 hours after drug administration